CLINICAL TRIAL: NCT00784030
Title: The Effect of Water Loading on Urinary Biomarkers
Brief Title: High Water Intake to Slow Progression of Polycystic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 08-774
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Results first posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Kidney, Polycystic, Autosomal Dominant
Keywords: Autosomal Dominant Polycystic Kidney Disease; Polycystic Kidney Disease; Water Loading; Biomarkers
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Polycystic Kidney Diseases | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polycystic Kidney Disease Patients (Other): Patients who present with polycystic kidney disease (PKD)
  Interventions: Other: Water
- Healthy Patients (Other)
  Interventions: Other: Water

INTERVENTIONS:
Other: Water — Participants will be first asked to drink 6 8-oz glasses of water over 2.5 hours on the first day, and then about 12 8-oz glasses of water over the course of the day for one week.

SUMMARY:
Polycystic kidney disease (PKD) is a genetic disease that occurs in 1 in 500 individuals and leads to kidney failure in half of all affected. Currently, no treatments exist for PKD. PKD-affected kidney cells divide and multiply inappropriately, and form fluid-filled sacs called cysts. Kidney cysts continue to grow throughout life, destroying normal kidney tissue, leading to kidney failure. Based on evidence from basic science research it is believed that drinking high amounts of water can slow the abnormal cysts growth. This study aims to look at changes in urine composition with high water intake in PKD-affected persons compared to healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Autosomal Dominant Polycystic Kidney Disease by history, ultrasound, CT or MRI
* Healthy subjects without a diagnosis of Polycystic Kidney Disease by history, ultrasound, CT or MRI
* Ages between 18 and 65
* Healthy subjects (without Polycystic Kidney Disease) must have an estimated glomerular filtration rate (eGFR by the MDRD equation) > 60 ml/min/1.73 m2 with no history of kidney disease

Exclusion Criteria:

* Women who are pregnant or nursing
* Active dependency on drugs or alcohol
* Diagnosis of syndrome of inappropriate antidiuresis
* Currently taking a vasopressin agonist or antagonist
* Blood sodium level less than < 135 mEq/L
* For healthy participants, estimated glomerular filtration rate (level of kidney function) less than < 60 ml/min/1.73 m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irina Barash, M.D., Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Polycystic Kidney Disease (PKD) Patients: Patients who present with polycystic kidney disease (PKD)
Period: Overall Study
Arm/Group | Polycystic Kidney Disease (PKD) Patients | Healthy Patients
Started | 13 | 10
Completed | 13 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polycystic Kidney Disease (PKD) Patients | Healthy Patients | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 10 | 23
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Urine cAMP Concentration and Urine Osmolality (UOsm)
Description: Urine cAMP (UcAMP) concentration and urine osmolality UOsm) were measured pre- and post-water loading: with 2.5L over 2 hours
Time Frame: pre- and post-water loading (2 hours)
Population: Number of participants was deemed to be adequate for the purposes of this pilot study
Measure: Mean (Standard Error); unit: fold change in cAMP/UOsm (umol/UOsm)
Groups:
- Polycystic Kidney Disease Patients: Patients with Autosomal Dominant Polycystic Kidney Disease
- Healthy Controls: Healthy Controls
Arm/Group | Polycystic Kidney Disease Patients | Healthy Controls
Number analyzed (Participants) | 13 | 10
fold change in cAMP/UOsm (umol/UOsm) | -2.6 (0.2) | -2.0 (0.1)

ADVERSE EVENTS:
Arm/Group | Polycystic Kidney Disease Patients | Healthy Controls
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/10
Other Adverse Events (participants affected / at risk) | 0/13 | 0/10

LIMITATIONS AND CAVEATS:
This was a very small study, so larger numbers are needed. Urine cAMP measurement as a surrogate of response to water treatment needs further validation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No